CLINICAL TRIAL: NCT06865092
Title: Comparison of Injectable Platelet-rich Fibrin, Titanium Platelet-rich Fibrin, and 0.8% Hyaluronic Acid Applications in Wound Healing After Gingivectomy and Gingivoplasty Operations: Randomized Controlled Clinical Study.
Brief Title: Comparison of I-PRF, T-PRF, and 0.8% Hyaluronic Acid Applications in Wound Healing After Gingivectomy.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Özlem SARAÇ ATAGÜN, Asst. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSATAGUN3
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Gingival Overgrowth
Keywords: Gingival Overgrowth; Hyaluronic Acid; I-PRF; T-PRF; Gingivectomy
MeSH Terms: conditions — Gingival Overgrowth | interventions — proliferation regulatory factors, human urine; Hyaluronic Acid; Control Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled, single-blind, prospective clinical study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- •I-PRF Group (Experimental): Following gingivectomy with the conventional method (#15 scalpel), I-PRF is applied to the wound site and covered with periodontal dressing.
  Interventions: Biological: injectable platelet-rich fibrin
- • T-PRF Group (Experimental): Following gingivectomy with the conventional method, T-PRF is applied to the wound site and covered with periodontal dressing.
  Interventions: Biological: titanium-prepared platelet-rich fibrin
- •HA Group (Experimental): Following gingivectomy with the conventional method, 0.8% HA (Gengigel; Ricerfarma, Milan, Italy) is applied to the wound site and covered with periodontal dressing.
  Interventions: Drug: Hyaluronic Acid (HA)
- •Control Group (Experimental): : Following gingivectomy with the conventional method, the wound site is covered only with periodontal dressing, without additional biomaterials.
  Interventions: Other: control group

INTERVENTIONS:
Biological: injectable platelet-rich fibrin — Blood samples were collected in two 10 ml plastic tubes without anticoagulant. The tubes were centrifuged for 3 min at 2500 rpm in a centrifuge device and i-prf was obtained.
  Other Names: i-prf
  Arms: •I-PRF Group
Biological: titanium-prepared platelet-rich fibrin — The blood was drawn into a 20 ml syringe and immediately divided into two sterile grade IV titanium tubes containing 10 ml of blood. The tubes were placed opposite each other and centrifuged at 2700 rpm for 12 minutes at room temperature and t-prf was obtained.
  Other Names: t-prf
  Arms: • T-PRF Group
Drug: Hyaluronic Acid (HA) — 0.8% hyaluronic acid (HA) gel (Gengigel) was applied to the wound sites.
  Other Names: HA; 0.8% HA
  Arms: •HA Group
Other: control group — Nothing has applied.
  Arms: •Control Group

SUMMARY:
Objectives: This study aimed to evaluate the effect of injectable platelet-rich fibrin (i-prf), titanium-prepared platelet-rich fibrin (t-prf), and 0.8% hyaluronic acid (HA) gel on clinical periodontal parameters, wound healing, patient comfort and satisfaction after gingivectomy and gingivoplasty procedures routinely performed in the treatment of chronic inflammatory gingival overgrowth.

Materials and methods: In this clinical study, 60 systemically healthy patients with chronic inflammatory gingival overgrowth were randomly assigned to i-prf (n=15), t-prf (n=15), 0.8% HA (n=15), or control (n=15) groups and treated with gingivectomy and gingivoplasty after initial periodontal treatment. Pain and burning scores were evaluated with VAS 7 days after the procedures. Surgical areas were stained with Mira-2 tone and evaluated in ImageJ. Wound healing was evaluated using the Landry, Turnbull, and Howley (LTH) index and H2O2 foaming test at 7, 14, 21, and 28 days after the procedure. Clinical periodontal parameters assessed at baseline and 3 weeks after initial periodontal treatment were reassessed at 28 days following gingivectomy and gingivoplasty.

DETAILED DESCRIPTION:
All patients diagnosed with chronic inflammatory gingival overgrowth based on clinical and radiological examinations underwent initial periodontal treatment (IPT) following baseline clinical periodontal assessments. Additionally, they received comprehensive oral hygiene instructions. After three weeks, patients were recalled for follow-up, and clinical periodontal parameters were re-evaluated. Gingivectomy and gingivoplasty surgery were planned.

Gingival growth was graded according to the following indices: The buccolingual aspect of gingival growth was classified according to the MB index (defined by Seymour and later modified by Miranda et al.) and the vertical aspect was classified according to the GOI index (defined by Angelopoulos and Goaz and later modified by Miller et al.). Patients presenting with a score greater than 0 in both indices were included in the study.

A total of four groups were planned in the study: one control group and three test groups.

* Test Group 1: Following gingivectomy with the conventional method (#15 scalpel), I-PRF is applied to the wound site and covered with periodontal dressing.
* Test Group 2: Following gingivectomy with the conventional method, T-PRF is applied to the wound site and covered with periodontal dressing.
* Test Group 3: Following gingivectomy with the conventional method, 0.8% HA (Gengigel; Ricerfarma, Milan, Italy) is applied to the wound site and covered with periodontal dressing.
* Control Group: Following gingivectomy with the conventional method, the wound site is covered only with periodontal dressing, without additional biomaterials.

Clinical periodontal parameters were evaluated at baseline (T0), after IPT (T1), and in the 1st month after gingivectomy and gingivoplasty (T2). The gingival index (GI; Loe and Silness GI), plaque index (PI; Turesky-Gilmore-Glickman modification of the Quigley-Hein PI), bleeding on probing index (BOP), and probing depth (PD) were recorded. Using a Williams periodontal probe, the GI, BOP, and PD were assessed at six sites per tooth (excluding the third molar): three sites on the buccal surface (disto-buccal/labial, mesio-buccal/labial, and mid-buccal/labial) and three sites on the lingual surface (disto-lingual/palatal, mesio-lingual/palatal, and mid-lingual/palatal).

Conventional gingivectomy and gingivoplasty procedures were performed under local infiltration anesthesia. A 45-degree inclined external bevel incision was made using a surgical scalpel (Carbon, No. 15) and a gingivectomy blade (Hu-Friedy 15/16, Chicago, USA), starting from the distal end of the incision line. The interdental area was shaped using an Orban knife (Hu-Friedy 1/2, Chicago, USA), and any remaining granulation tissue was carefully removed from the surrounding area with curettes and scissors (Hu-Friedy, Chicago, USA). Finally, gingivoplasty was completed using a Kirkland knife (Hu-Friedy, Chicago, USA).

After the surgical procedures were completed, the control group areas were left to heal spontaneously. The other groups were treated with i-prf, t-prf, or 0.8% HA. Surgical areas in the control and test sites were covered with periodontal dressing (Coepak, Isip, IL, USA).

Patients were advised to avoid hot foods, to consume soft foods, and to keep the dressing in the mouth until the next examination. Patients were prescribed mouthwash containing 0.12% chlorhexidine and analgesic containing paracetamol to be used twice a day for one week.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18-65 years of age
2. Being systemically healthy
3. Having chronic inflammatory gingival overgrowth in the mandibular and maxillary anterior region, with no attachment and bone loss
4. Not to have used any medication in the last three months
5. Not smoking
6. At least 20 natural teeth

Exclusion Criteria:

1. Patients with orthodontic appliances
2. Patients with removable (partial) prostheses
3. Patients with immunosuppressive agents, systemic corticosteroids, chemotherapy, and/or radiotherapy drugs and/or drugs that may cause gingival enlargement use in the last 6 months
4. Patients with oral and/or peri-oral pain
5. Patients with significant oral lesions
6. Patients with antibiotic use in the last 3 months, pregnancy and breastfeeding
7. Patients who have undergone periodontal treatment within the last 6 months
8. Patients with poor communication skills
9. Smokers and alcohol users

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of wound epithelialization | after gingivectomy (Day 0), Day 7, Day 14, Day 21, Day 28
  Evaluation of wound epithelialization with Mira-2 tone Solution
LTH wound healing index | Day 7, Day 14, Day 21, Day 28
  Assessment of soft tissue healing with Landry, Turnbull, and Howley (LTH) index

SECONDARY OUTCOMES:
H2O2 foaming test | Day 7, Day 14, Day 21, Day 28
  H2O2 foaming test (evaluation of wound epithelialization)
Pain and burning scores | After gingivectomy Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
  Pain and burning scores were evaluated with VAS.
Gingival index (GI) | Baseline, 3 weeks, Day 28 after gingivectomy
  Improvement in GI; lower scores mean a better outcome; Minimum score:0 Max.score: 3
Plaque index (PI) | Baseline, 3 weeks, Day 28 after gingivectomy
  Improvement in PI; lower scores mean a better outcome; Minimum score:0 Max.score: 5
Bleeding on Probing (BOP) | Baseline, 3 weeks, Day 28 after gingivectomy
  Improvement in PBI; lower scores mean a better outcome; Minimum score: %0 Max.score: %100
Pocket depth (PD) | Baseline, 3 weeks, Day 28 after gingivectomy
  Improvement in PD; lower scores mean a better outcome
OHIP-14 | Baseline, Day 7, Day 14 after gingivectomy
  Improvement in Oral Health Impact Profile (OHIP-14) ; lower scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: özlem saraç atagün, PhD, Principal Investigator — Sağlık Bilimleri Üniversitesi Gülhane Diş Hekimliği Fakültesi Periodontoloji AD
Locations (1):
- Sağlık Bilimleri Üniversitesi Gülhane Diş Hekimliği Fakültesi, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No